CLINICAL TRIAL: NCT03716570
Title: A Multicenter, Blinded, Placebo-Controlled, Randomized, Single and Multiple-Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BIIB054 in Japanese Subjects With Parkinson's Disease
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BIIB054 in Japanese Participants With Parkinson's Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Affiliated study NCT03318523 did not meet its primary outcome measure of change from baseline measured by Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) and did not demonstrate efficacy on secondary outcome measures
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 228PD103
Record Dates: First submitted 2018-10-22; First posted 2018-10-23 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1: BIIB054 Dose A (Experimental): Participants will receive IV infusion of BIIB054 Dose A (single infusion on Day 1 followed by an observation period; with subsequent doses for 48 weeks)
  Interventions: Drug: BIIB054
- Cohort 2: BIIB054 Dose B (Experimental): Participants will receive IV infusion of BIIB054 Dose B (single infusion on Day 1 followed by an observation period; with subsequent doses for 48 weeks)
  Interventions: Drug: BIIB054
- Cohort 3: BIIB054 Dose C (Experimental): Participants will receive IV infusion of BIIB054 Dose C (single infusion on Day 1 followed by an observation period; with subsequent doses for 48 weeks)
  Interventions: Drug: BIIB054
- Cohorts 1-3: Placebo (Placebo Comparator): Participants will receive a single IV infusion of BIIB054 matching placebo (single infusion on Day 1 followed by an observation period; with subsequent doses for 48 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB054 — Administered as specified in the treatment arm.
  Arms: Cohort 1: BIIB054 Dose A; Cohort 2: BIIB054 Dose B; Cohort 3: BIIB054 Dose C
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Cohorts 1-3: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of a range of single and 13 repeated doses of BIIB054, administered as intravenous (IV) infusion, in Japanese participants with Parkinson's disease (PD). The secondary objectives are to evaluate the immunogenicity, and serum pharmacokinetics (PK) profile of BIIB054 after single and multiple dose administration.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with PD within a maximum of 3 years prior to screening.
* Has not received levodopa or any other treatment for PD, herein referred to as symptomatic PD medication (including but, not limited to, dopamine agonists, amantadine, anticholinergics, monoamine oxidase type B (MAO-B) inhibitors, or safinamide) for at least 12 weeks prior to Day 1. Maximum total duration of prior PD regimens should not exceed 30 days.
* Score of less than equal to (<=) 2.5 on the Modified Hoehn and Yahr Scale.
* Screening dopamine transporter (DaT)/ single-photon emission computed tomography (SPECT) results consistent with neurodegenerative Parkinsonism (central reader).

Key Exclusion Criteria:

* Presence of freezing of gait.
* History of or positive test result at Screening for human immunodeficiency virus (HIV) or hepatitis C virus antibody (anti-HCV).
* Screening value for hemoglobin less than (<)12 gram per deciliter (g/dL) for men or <11 g/dL for women.
* Montreal Cognitive Assessment (MoCA) score <23 or other significant cognitive impairment or clinical dementia.
* History of any brain surgery for PD.
* Participation in any passive or active immunotherapy targeting alpha-synuclein or other PD-related protein.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 72 Weeks
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death, is a life-threatening event, requires inpatient hospitalization or prolongation of existing hospitalization, results in a significant disability/incapacity or congenital anomaly, or is a medically important event.

SECONDARY OUTCOMES:
Area Under the Serum Concentration-Time Curve From Time Zero Extrapolated to Infinite Time (AUCinf) of BIIB054 | Up to 24 Weeks
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of BIIB054 | Up to 24 Weeks
Maximum Observed Serum Concentration (Cmax) of BIIB054 | Up to 24 Weeks
Time to Reach Maximum Observed Serum Concentration (Tmax) of BIIB054 | Up to 24 Weeks
Terminal Elimination Half-life (t1/2) of BIIB054 | Up to 24 Weeks
Clearance (CL) of BIIB054 | Up to 24 Weeks
Volume of Distribution at Steady State (Vss) of BIIB054 | Up to 24 Weeks
Accumulation Ratio of BIIB054 | Up to 24 Weeks
Observed Concentration at the End of Dosing Interval (Ctrough) of BIIB054 | Up to 24 Weeks
Number of Participants With Anti-BIIB054 Antibodies in Serum | Up to 72 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (7):
- Japan (7):
  - Research Site, Toon-shi, Ehime
  - Research Site, Asahikawa-shi, Hokkaido
  - Research Site, Kyoto, Kyoto
  - Research Site, Sendai, Miyagi
  - Research Site, Suita-shi, Osaka
  - Research Site, Bunkyō City, Tokyo-To
  - Research Site, Kodaira-shi, Tokyo-To

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/

REFERENCES:
- See also: Fox Trial Finder — https://foxtrialfinder.michaeljfox.org/trial/6140